CLINICAL TRIAL: NCT05238155
Title: Evaluation of the Impact of Reduced Immunosuppression on Graft-versus-host Disease and Rejection Rates in Orthotopic Liver Transplant Recipients
Brief Title: Evaluation of the Impact of Reduced Immunosuppression
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 041.PHA.2021.D
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Antimetabolites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthotopic Liver Transplantation recipients prior to protocol implementation date: Orthotopic Liver Transplantation recipients are discharged following transplantation, they are typically prescribed a triple immunosuppression maintenance regimen, consisting of a calcineurin inhibitor, an antimetabolite, and a corticosteroid.
  Interventions: Drug: antimetabolite
- Orthotopic Liver Transplantation recipients after protocol implementation date: Over the last several years, there have been changes made to this protocol, and the current protocol now suggests consideration for the omission of the antimetabolite at discharge if there is a donor-recipient age discrepancy that is greater than 30 years. This change was made with the intention to reduce the risk of GVHD, given that a greater disparity in donor-recipient age may put these patients at a higher risk for GVHD.

INTERVENTIONS:
Drug: antimetabolite — When OLT recipients are discharged following transplantation, they are typically prescribed a triple immunosuppression maintenance regimen, consisting of a calcineurin inhibitor, an antimetabolite, and a corticosteroid. Over the last several years, there have been changes made to this protocol, and the current protocol now suggests
  Groups: Orthotopic Liver Transplantation recipients prior to protocol implementation date

SUMMARY:
Graft-versus-host disease (GVHD) is a life-threatening complication of transplantation. It occurs when the donor graft contains immunologically competent T-cells that recognize the recipient as foreign.

DETAILED DESCRIPTION:
GVHD is commonly observed in allogeneic hematopoietic stem cell transplantation recipients but can also occur in recipients of solid organ transplantation , with the first case of GVHD in a SOT recipient described in 1984. While the exact incidence of SOT-associated GVHD has not been determined due to challenges with identifying and diagnosing GVHD in SOT recipients, the reported incidence of GVHD following orthotopic liver transplantation ranges from 0.1%-2%, one of the highest rates among SOT recipients. Although it occurs very rarely with SOT, GVHD leads to poor patient outcomes, with a mortality rate exceeding 75%. Risk factors for SOT-associated GVHD have not been clearly defined, but possible risk factors have been identified, such as recipient age ≥65 years, donor-recipient age difference of ≥40 years, degree of human leukocyte antigen matching, level of immunosuppression, and history of hepatocellular carcinoma.

There are currently no guideline recommendations for treatment or prevention of GVHD in SOT patients. Current treatment strategies include a combination of increasing immunosuppression, decreasing immunosuppression, or changing immunosuppression agents, making it difficult to definitively determine an effective treatment approach.

However, it has been postulated that decreasing immunosuppression may allow the transplant recipient's native immune system to reject donor lymphocytes and would therefore act protectively against GVHD in these patients. Since there is currently no clinical outcomes data to support this and because GVHD is a very rare occurrence in this population, reducing immunosuppression as a preventative measure for GVHD is not a commonplace practice amongst SOT centers.

The Liver Institute at Methodist Dallas Medical Center (MDMC) is a comprehensive, multidisciplinary disease management center. One of its services is OLT with life-long outpatient follow-up. When OLT recipients are discharged following transplantation, they are typically prescribed a triple immunosuppression maintenance regimen, consisting of a calcineurin inhibitor, an antimetabolite, and a corticosteroid. Over the last several years, there have been changes made to this protocol, and the current protocol now suggests consideration for the omission of the antimetabolite at discharge if there is a donor-recipient age discrepancy (DAD) that is greater than 30 years. This change was made with the intention to reduce the risk of GVHD, given that a greater disparity in donor-recipient age may put these patients at a higher risk for GVHD.

Since this protocol implementation, the exact clinical implications of this reduction in immunosuppression are still unclear. While this approach may reduce the incidence of GVHD, omission of the antimetabolite in maintenance immunosuppression regimens puts these OLT recipients at risk for rejection of their graft, which can also be a life-threatening complication. Evaluation of the clinical outcomes related to this protocol change is warranted in order to appropriately weigh the risks versus benefits of reducing immunosuppression to prevent GVHD.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Received OLT or CKLT during study period

Exclusion Criteria:

* Recipients requiring re-transplant within one month post-transplant
* Recipients who died of a cause other than GVHD within one month post-transplant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients admitted for OLT or combined kidney-liver transplant
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-10-19 (Estimated); Study Completion 2024-10-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of GVHD at one year post-transplant | September 12, 2004 to June 30, 2020
  Diagnosis confirmed with donor lymphoid chimerism
Graft rejection at one year post-transplant | September 12, 2004 to June 30, 2020
  Diagnosis confirmed by liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Crotty, PharmD, Principal Investigator — Methodist Health System
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No